CLINICAL TRIAL: NCT00227669
Title: Randomized Phase II Study Evaluating the Efficacy of Gemcitabine Versus the Gemcitabine/Docetaxel Combination as Second Line Treatment in Metastatic or Relapsed and Inoperable Uterine or Soft Tissue Leiomyosarcomas
Brief Title: Gemcitabine With or Without Docetaxel as Second-Line Therapy in Treating Patients With Metastatic or Relapsed, Unresectable Uterine or Soft Tissue Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000443572; FRE-FNCLCC-SARCOME-07/0410; EU-20518
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Sarcoma
Keywords: uterine leiomyosarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; adult leiomyosarcoma
MeSH Terms: conditions — Sarcoma; Leiomyosarcoma | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Gemcitabine (Active Comparator): Gemcitabine at Day 1, Day 8 and Day 15. No treatment at Day 22.
  1 cycle = 28 days.
  Treatment duration: 8 months
  Interventions: Drug: gemcitabine hydrochloride
- Arm II: Gemcitabine + Docetaxel (Experimental): Gemcitabine at Day 1 and Day 8. No treatment at Day 15. Docetaxel at Day 8.
  1 cycle = 21 days.
  Treatment duration: 6 months
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: docetaxel
  Arms: Arm II: Gemcitabine + Docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether giving gemcitabine together with docetaxel is more effective than giving gemcitabine alone as second-line therapy in treating uterine or soft tissue leiomyosarcoma.

PURPOSE: This randomized phase II trial is studying gemcitabine and docetaxel to see how well they work compared to gemcitabine alone as second-line therapy in treating patients with metastatic or relapsed, unresectable uterine or soft tissue leiomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the anti-tumor activity, in terms of objective response rate, in patients with metastatic or relapsed, unresectable uterine or soft tissue leiomyosarcoma treated with gemcitabine with vs without docetaxel as second-line therapy.

Secondary

* Compare the progression-free survival of patients treated with these regimens.
* Compare the response duration and overall survival of patients treated with these regimens.
* Compare the tolerability and dose intensity of these regimens in these patients.
* Determine biological markers with a predictive value for response to these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to location of leiomyosarcoma (uterine vs soft tissue). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine on days 1, 8, and 15. Treatment repeats every 4 weeks for 2-8 courses.
* Arm II: Patients receive gemcitabine on days 1 and 8 and docetaxel on day 8. Treatment repeats every 3 weeks for 2-8 courses.

PROJECTED ACCRUAL: A minimum of 80 patients (40 per stratum and treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed uterine or soft tissue leiomyosarcoma, meeting ≥ 1 of the following criteria:

  * Metastatic disease
  * Relapsed and unresectable disease
* Prior treatment with a first-line anthracycline-based chemotherapy regimen required

  * Relapsed disease > 1 year after adjuvant chemotherapy is considered untreated disease
  * If relapsed disease occurs < 1 year after adjuvant therapy, then adjuvant therapy is considered a first-line treatment
* At least 1 measurable lesion, defined as the following:

  * At least 1 target lesion must be located in a non-irradiated area
  * Obvious disease progression within the past 6 weeks
* No other uterine sarcomas, including any of the following:

  * Carcinosarcoma
  * Endometrial stroma sarcoma
  * Other soft tissue sarcoma
* No symptomatic or known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* No specific hepatic contraindication to study treatment
* Hepatitis B core and hepatitis B surface antigen negative

Renal

* Creatinine < 1.5 times ULN
* No specific renal contraindication to study treatment

Cardiovascular

* No specific cardiac contraindication to study treatment

Immunologic

* HIV negative
* No specific allergic contraindication to study treatment
* No active infection

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other serious underlying pathology that would preclude study treatment
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No neurotoxicity > grade 2
* No psychological, sociological, or geographical condition that would preclude study compliance or follow-up schedule
* No prior or concurrent psychiatric illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* No prior allogeneic graft or autologous graft

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy
* No prior gemcitabine and/or taxane (i.e., docetaxel or paclitaxel)

Endocrine therapy

* More than 4 weeks since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to the only evaluable lesion

Surgery

* Not specified

Other

* No concurrent participation in another clinical trial using an experimental agent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-10; Primary Completion 2010-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Anti-tumoral activity (objective response rate) | 6 months

SECONDARY OUTCOMES:
Progression-free survival | 6 months
Response duration | 3 years
Tolerability | 3 years
Dose intensity | 3 years
Overall survival | 3 years
Biological markers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Florence Duffaud, MD, Study Chair — CHU de la Timone
Locations (32):
- France (32):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Centre Paul Papin, Angers
  - C.H.G. Beauvais, Beauvais
  - Institut Bergonie, Bordeaux
  - C.H.U. de Brest, Brest
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - CHU de la Timone, Marseille
  - CHU Nord, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Bichat - Claude Bernard, Paris
  - Institut Curie Hopital, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Cochin, Paris
  - CHU Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Hopital Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared at an individual level.

REFERENCES:
- [Result] Duffaud F, Bui BN, Penel N, et al.: A FNCLCC French Sarcoma Group--GETO multicenter randomized phase II study of gemcitabine (G) versus gemcitabine and docetaxel (G+D) in patients with metastatic or relapsed leiomyosarcoma (LMS). [Abstract] J Clin Oncol 26 (Suppl 15): A-10511, 2008.